CLINICAL TRIAL: NCT06935747
Title: Clinical Study to Analyze the Osteogenic Action of a Beta-tricalcium Phosphate-based Product in Bone Regeneration After the Extraction of Impacted Mandibular Third Molars.
Brief Title: Osteogenic Action of a Medical Device Based on Beta-tricalcium Phosphate (BTCP)
Acronym: BTCP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Pérez Sayáns (Other)
Collaborators: Universidad de Murcia (Other); Nueva Galimplant SLU (Unknown)
Responsible Party: Sponsor-Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Organization: University of Santiago de Compostela (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTCP2025
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Bone Loss; Regenerative Inflammation; Third Molars Extraction
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BTCP Group (Experimental): The experimental BTCP group includes participants who will receive BTCP after the extraction of an impacted mandibular third molar to test its osteogenic properties. BTCP is prepared according to the manufacturer's instructions, initially by immersing it in sterile saline solution. It is applied to the socket after extraction using specialized instruments and is compared with a control group that receives Bio-Oss, a standard xenograft material.
  Patients in the experimental group receive postoperative medication, including antibiotics and pain management treatment. Follow-up evaluations assess pain, inflammation, complications, and bone regeneration through radiological assessment.
  Objective: To evaluate the efficacy of BTCP in bone regeneration compared to the control.
  Interventions: Combination Product: Medical device: beta-tricalcium phosphate
- Control group (Active Comparator): The control group serves as the active comparator to the BTCP experimental group in this study. Participants undergo the same impacted mandibular third molar extraction procedures as those in the experimental group, but receive a standard material, Bio-Oss, instead of BTCP.
  Bio-Oss, a widely used xenograft material in dental surgeries, serves as the reference due to its osteoconductive properties. It is applied to the socket after extraction using specialized instruments and acts as a benchmark for comparing the efficacy of BTCP. Patients in the control group receive postoperative medication according to the study protocol, including antibiotics and pain management treatment. Follow-up assessments evaluate pain, inflammation, complications, and bone regeneration through radiological evaluation.
  Interventions: Other: Bovine Hydroxyapatite

INTERVENTIONS:
Combination Product: Medical device: beta-tricalcium phosphate — The description of the intervention for BTCP in the study involves the application of this substance to promote bone regeneration following the extraction of impacted mandibular third molars. BTCP is indicated for the treatment of segmental and cavitary bone loss, aesthetic repairs, and bone augmentations (such as inlay or onlay grafts); for filling dental alveolar bone; for dental implant placement; and for the stabilization of osteotomies and prostheses in dentistry.
  Arms: BTCP Group
Other: Bovine Hydroxyapatite — The intervention description for Bio-Oss in the study involves the application of this standard material to promote bone regeneration following the extraction of impacted mandibular third molars. Bio-Oss is a commonly used xenograft material known for its osteoconductive properties.
  Arms: Control group

SUMMARY:
The general objective of this split-mouth study is to analyze the osteogenic action of BTCP during the bone regeneration process following the extraction of impacted mandibular third molars.

DETAILED DESCRIPTION:
The proposed protocol is a multicenter clinical trial aimed at analyzing the osteogenic action of a medical device based on beta-tricalcium phosphate (hereinafter BTCP) in the bone regeneration process following the extraction of impacted mandibular third molars. The specific objectives of the study include a comparative analysis of clinical and radiological variables between a control group and a study group.

Inclusion criteria for study subjects include being of legal age, providing informed consent, and requiring the extraction of both impacted mandibular third molars, among others. Exclusion criteria include the presence of severe mental disorders or medical contraindications for tooth extraction.

The study involves a total of 60 third molars from 30 patients, divided into a control group and a study group. Data will be collected regarding patient demographics, the surgical procedure, and the bone regeneration assessment.

The surgical procedure involves selecting patients with similarly complex third molars, followed by tooth extraction and the placement of BTCP in the study group or a standard material in the control group. Clinical follow-up will be conducted during the first 7 days, and radiological follow-up will take place over the following 6 months to evaluate bone regeneration.

Patients will receive compensation for their participation in the study, which includes medical consultations, phone follow-ups, examination time, completion of questionnaires, and training in self-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be of legal age, generally defined as 18 years or older, to be able to provide adequate informed consent and understand the risks and benefits of the procedure.
* Informed Consent: Patients must be willing to provide written informed consent to participate in the study, indicating their understanding and acceptance of the associated procedures and risks.
* Need for Extraction of Impacted Mandibular Third Molars: Patients must require the extraction of both impacted mandibular third molars to be eligible for the study.
* Similar Complexity of Impacted Third Molars: The impacted mandibular third molars must present similar complexity for extraction on both sides of the jaw, to ensure a fair comparison between the study groups.
* Absence of Medical Contraindications for Oral Surgical Procedures: Patients must not have significant medical contraindications that would prevent oral surgical procedures, such as clotting disorders, uncontrolled systemic diseases, or a history of severe infections.

Exclusion Criteria:

* Severe Mental Disorders: Patients with severe mental disorders that may affect their ability to understand and follow study instructions may be excluded due to concerns about their capacity to provide valid informed consent and follow the study protocol.
* Contraindications for Dental Extractions: Patients with specific contraindications for dental extraction, such as a history of osteonecrosis of the jaws or serious complications associated with previous dental procedures, may be excluded for safety reasons.
* Patients under the age of 18 will not be eligible to participate in the study due to ethical and legal concerns related to obtaining informed consent and the ability to understand the risks and benefits of the study.

Withdrawal from the Study:

-If a patient experiences severe complications during the study, such as severe postoperative infections, severe allergic reactions, or any other adverse event that may jeopardize their health, they will be considered for withdrawal from the study to ensure their well-being. Additionally, if a patient decides to voluntarily withdraw from the study at any time, their decision will be respected, and appropriate medical care will be provided as needed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Bone Regeneration_Reduction in radiolucent volume | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction. Reduction in radiolucent volume within the extraction socket, indicating new bone formation (Hounsfield unit (HU)). High values mean more radiopacity and better regeneration.
Bone Regeneration_bone volume | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction. Evaluation of bone volume within the extraction site over time (mm3). The increase in bone volume means better regeneration
Bone Regeneration_bone density | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction. Changes in bone density within the regenerated bone tissue (Hounsfield unit (HU)) High values mean more radiopacity and better regeneration.
Bone Regeneration_Fractal dimension | A) Immediately after extraction B) 1 month. C) 3 months. D) 6 months
  This outcome measure involves assessing the degree of bone regeneration in the extraction socket following the extraction of impacted mandibular third molars. It will be evaluated through radiological imaging using CBCT scans at specified time points, including immediately post-extraction, at one month, three months, and six months post-extraction. Evaluation of bone morphology within the extraction site over time analyzing the fractal dimension (FD) FD can vary between 1 and 2, with 1 being a very simple fractal dimension (such as a straight line) and 2 being a more complex fractal dimension (such as a completely irregular surface)

SECONDARY OUTCOMES:
Pain levels through visual analog scale | 24 hours, 48 hours, 72 hours, and 7 days
  Assessment of pain experienced by participants using a visual analog scale (VAS) at various time points post-extraction. It comprehends values between 0-10, where 10 is the worst situation.
Clinical Inflammation evaluating by presence/absence | 24 hours, 48 hours, 72 hours, and 7 days
  Evaluation of postoperative inflammation around the extraction site using clinical examination and assessment tools (presence/absence). The presence of inflammation means the worst prognosis.
Healing measured by healing index | 24 hours, 48 hours, 72 hours, and 7 days
  The healing progress will be assessed using the Healing Index (HI) developed by Hamzani & Chaushu (2018) and Landry (1988). The HI score ranges from 0 to 5, where 0 indicates poor healing and 5 indicates excellent healing. To ensure consistency and reliability in the assessment of healing, two independent researchers will evaluate the healing progress for all participants. The level of agreement between the researchers will be assessed using Cohen's Kappa index (Mandrekar, 2011). A Cohen's Kappa index value of 0.91 was achieved for the assessment of inflammation level, indicating a high degree of agreement. Similarly, agreement levels exceeding 0.90 were obtained across all HI levels, demonstrating a high level of concordance in the assessment of healing progress.
Post-surgical complications evaluated by presence or absense | 24 hours, 48 hours, 72 hours, and 7 days
  Monitoring and recording of any complications following the extraction procedure, such as alveolitis, trismus, infection, and hematoma (presence/absence). The presence of complications is related to a worse prognosis.
Oral Health-related Quality of Life measured by OHIP-14 test | 24 hours, 48 hours, 72 hours, and 7 days
  Assessment of the impact of treatment on patients' quality of life using validated instruments (OHIP-14). The higher the average value of the seven dimensions, the more negative the impact of oral health on the quality of life of an individual.Minimum of 0 points and maximum of 56 points. Lower scores: They indicate that the person experiences less impact of oral health problems on their quality of life. That is, they have fewer problems or feel less the impact of these problems in their daily lives. Intermediate scores: Suggest a moderate impact of oral health problems on quality of life. The person may experience some difficulties or discomfort related to their oral health, but they do not necessarily significantly affect their daily functioning. Higher scores: Indicate a significant impact of oral health problems on quality of life. The person may experience a wide range of problems that affect their general well-being, including pain, eating difficulties, sleep problems, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Camacho Alonso, phD, Principal Investigator — Universidad de Murcia; Abel García García, phD, Study Chair — Universidade de Santiago de Compostela
Locations (2):
- Spain (2):
  - Universidade de Santiago de Compostela, Santiago de Compostela, A Coruña
  - University of Murcia, Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No